CLINICAL TRIAL: NCT06601712
Title: Delivery Strategies for Malaria Chemoprevention in the Post-discharge Management of Children Hospitalised With Severe Anaemia or Severe Malaria: a Cluster Randomised Controlled Implementation Trial in Benin
Brief Title: Post-discharge Malaria Chemoprevention Implementation Trial in Benin
Acronym: PDMC-SL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Institut de Recherche Clinique du Benin (Other)
Collaborators: Liverpool School of Tropical Medicine (Other); Kenya Medical Research Institute (Other); Epicentre, Paris, France and Mbarara University of Science and Technology, Faculty of Medicine, Mbarara, Uganda (Other); Institut de Recherche pour le Developpement (Other Government); Training Research Unit of Excellence, Blantyre, Malawia (Unknown); Centres for Disease Control and Prevention, Kenya. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 191-20231218
Record Dates: First submitted 2024-08-13; First posted 2024-09-19 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Severe Malaria; Severe Anaemia
Keywords: Children; Antimalarial; Prevention; Chemoprevention; Caregivers; Patient discharge; Health care providers; Health economics; Qualitative research; Feasibility; Cost-effectiveness; Benin; Artemisinins; School age; Pre-school
MeSH Terms: conditions — Malaria; Anemia

STUDY DESIGN:
Intervention Model Description: A multi-centre cluster randomized implementation trial with three arms at health facilities and their catchment communities (clusters) to enhance end-user adherence to post-discharge malaria chemoprevention (PDMC) compared to a control arm of PDMC without specific adherence support strategies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): All PDMC drugs will be given to the caregivers at discharge with reminder support
  Interventions: Other: Adherence support strategy A
- Arm B (Experimental): All PDMC drugs will be given by the community health workers (CHWs) to the caregivers at home, with reminder support
  Interventions: Other: Adherence support strategy B
- Arm C (Active Comparator): All PDMC drugs will be given to the caregivers at discharge with no other adherence support approaches (no reminder)
  Interventions: Other: Control

INTERVENTIONS:
Other: Adherence support strategy A — Community health worker (CHW) support through monthly home visits to remind the caregiver to administrate the PDMC drugs
  Arms: Arm A
Other: Adherence support strategy B — SMS/phone reminders from the qualified community health officers (ASCQ) to the community health workers (CHW) to administrate the PDMC drugs
  Arms: Arm B
Other: Control — No reminders
  Arms: Arm C

SUMMARY:
The proposed research aims to conduct implementation trials in Benin, co-designed with national stakeholders, to evaluate different delivery strategies for optimizing health system delivery of post-discharge malaria chemoprevention (PDMC) drugs and adherence to PDMC. This chemoprevention strategy is effective in reducing hospital readmissions and deaths after discharge. However, there is no clear delivery platform for PDMC, and adherence to the 3-day dosing regimen, provided monthly three times after discharge, is a potential limitation. The current trial will provide evidence-based data on acceptability, feasibility, and cost-effectiveness to aid decision-makers. The evidence generated will be used to support the effective implementation and scale-up of PDMC in high malaria-endemic areas such as Benin.

DETAILED DESCRIPTION:
Introduction : Severe anaemia is a major cause of morbidity and mortality in children in malaria-endemic areas of sub-Saharan Africa, accounting for a large fraction of paediatric hospitalisations and in-hospital mortality [1] However, these children also remain at high risk of dying or being readmitted after discharge from hospital due to a wide range of clinical, epidemiological, behavioural and nutritional factors [2,3]. A recent trial in East Africa showed that about a third of discharged children after recovery from severe anaemia were readmitted or died in the first 6 months post-discharge [4]. In highly endemic settings, malaria is a major cause of this post-discharge morbidity and mortality [5,6].

In June 2022, the World Health Organization (WHO) recommended PDMC for the post-discharge management of children with severe anaemia in settings with moderate to high perennial malaria transmission to reduce hospital readmissions and deaths after discharge [7,8]. However, there is no obvious delivery platform for PDMC, unlike for intermittent preventive treatment in infants (IPTi) or pregnant women (IPTp). Furthermore, a potential limitation of PDMC is adherence to the 3-day dosing regimen, which is provided monthly three times after discharge. Therefore, implementation research is urgently needed to support the introduction and scale-up of PDMC. We propose to conduct two implementation trials to evaluate delivery strategies to optimise adherence to PDMC in different contexts: one in East Africa (Kenya) and one in West Africa (Benin). The current protocol presents the trial description in Benin.

Rationale of the trial: The WHO recommendation highlighted the need for implementation research on optimal delivery strategies for PDMC to help guide decision-making. The WHO recommendation stopped short of recommending which antimalarial drug should be used and how best to deliver PDMC, indicating that these decisions are to be made at the national level and adapted to suit local contexts. Importantly, the recommendation does not recommend any one specific drug or regimen to be used for PDMC, stating "SP, AL and DP were used in three trials and all regimens were found to be effective for PDMC" and "the medicines used for PDMC can be the same as the first-line malaria treatment, but an alternative medicine is preferred". Neither does the recommendation provide guidance on the optimal delivery mechanism(s) for giving the post-discharge chemoprevention regimen to caregivers in a way that promotes adherence and public health impact. A major challenge with implementing PDMC is that there is no pre-existing platform that could be utilised for its delivery. This is in contrast to other malaria prevention strategies, such as seasonal malaria chemoprevention (SMC), intermittent preventive treatment in pregnant women (IPTp), and perennial malaria chemoprevention (PMC, previously known as IPTi) and the recently recommended RTS,S malaria vaccine. Currently, the evidence on how to implement PDMC is limited to a single implementation trial in Malawi [8]. Furthermore, it must be appreciated that health systems, particularly in the community, vary from country to country. The adherence to monthly 3-day courses of PDMC after discharge under real-life conditions is unknown.

Study objectives:

The primary objective is to determine the effectiveness of different community delivery mechanisms and adherence support strategies to optimise end-user adherence to PDMC. Secondary objectives are to: i) determine the clinical effectiveness of the different PDMC delivery strategies (all-cause and malaria-specific readmissions and sick-child clinic visits, all-cause mortality); ii) evaluate the effectiveness of the linkage mechanisms between the various health facility levels along the PDMC delivery continuum; iii) determine the acceptability and feasibility of the different PDMC delivery and adherence support strategies; iv) determine the incremental cost-effectiveness (cost per DALY averted) of the different PDMC delivery and adherence support strategies.

Study design: The trial is a cluster randomized implementation trial with three arms at health facilities and their catchment communities (clusters) to enhance end-user adherence to the three PDMC courses compared to a control arm of PDMC without specific adherence support strategies. Its goal is to translate PDMC research findings into national policy guidelines and encourage their adoption in clinical practice, ensuring that caregivers of vulnerable children in Benin, and more broadly across sub-Saharan Africa, gain access to life-saving, proven medicines that help prevent or reduce hospital readmissions and deaths.

Study sites: Two health facilities with blood transfusion services will include in the trial in Benin. The recruitment will be competitive between the two selected hospitals over approximately 14 months to reach the study sample size. The first site, CHU-MEL has a higher annual incidence of severe anaemia (approximately 800-1000 cases per year) than the second site, Goho departmental hospital centre. Therefore, the proportion of participants enrolled at CHU-MEL could be slightly higher than in Goho.

Study population:

Inclusion criteria: convalescent children aged below 10 years, weighing above or equal to 5 kg admitted with severe anaemia (haemoglobin below 5g/dL) or severe malaria; clinically stable, able to take or switch to oral medication; post-transfusion Hb below 5g/dL.

Exclusion criteria: blood loss due to trauma, malignancy, known bleeding disorders or sickle cell disease, known hypersensitivity to study drug, known heart conditions, non-resident in the study area, previous participation in the study, known need at enrolment for prohibited medication and scheduled surgery during the 6-month course of the study. HIV infection and cotrimoxazole prophylaxis are not exclusion criteria.

Study intervention: The final choice of drug, the delivery strategy and the adherence support mechanisms to be evaluated have been co-designed with MoH and key national public health stakeholders through formative research conducted under a separate standalone protocol and through a stakeholder co-design workshop. In Benin, PDMC will comprise of 3-day treatment courses either dihydroartemisinin-piperaquine given at the end of weeks 2, 6, and 10 after discharge. PDMC will consist of three courses of dihydroartemisinin-piperaquine at the end of weeks 2, 6, and 10 after discharge.

Two community delivery strategies combined with adherence supports will be assessed during the trial: (i) all the drugs given at discharge to the caregivers (strategy A); (ii) all the drugs will be given by the community health workers (CHWs) to the caregivers at home, supervised by the qualified community health officers (ASCQ) (strategy B). Clusters will be randomly allocated in a 1:1:1 ratio to intervention (a, b) and the control (c) arms. The unit of randomization will be health facilities's catchment villages to avoid contamination related to adherence supports in community. Each health facility and its respective community will form a cluster. In arm "a", all PDMC drugs will be given to the caregivers at discharge with the CHW support through monthly home visits to remind the caregiver to administrate the PDMC drugs; and in arm "b" all PDMC drugs will be given by the community health workers (CHWs) to the caregivers at home, with a SMS/phone reminder from the qualified community health officers (ASCQ). Arm "c" represents the control arm (no reminder), in which all PDMC drug given to the caregivers at discharge with no other adherence support approaches.

All participating children will receive standard in-hospital care for severe anaemia or severe malaria (blood transfusion, often combined parenteral artesunate, followed by a 3-day course of artemether-lumefantrin (whether they initially had malaria or not), which will be started in-hospital as soon as they are able to take oral medication. Many children are likely to receive parenteral antibiotics as well as part of the standard of care.

Economic evaluation: The cost of delivering the intervention from the providers perspective and the cost of receiving the intervention from the beneficiary's perspective will be assessed through an economic evaluation (cost-effectiveness analysis) involving all children (and their caregivers) participating in the trials in both countries. The same participant groups included in the acceptability and feasibility study, as well as hospital and peripheral facility managers, health workers responsible for the delivery of PDMC interventions (including community health workers) will be requested to support the provider costing. Malaria control programme managers, other regional, national and international stakeholders will be requested to provide perspectives on how PDMC could integrate with existing general health and malaria budget structures, and the size and flexibility of relevant budgets. This information will be used to inform a budget impact assessment of scaling up PDMC.

Acceptability and feasibility: A health services qualitative study will be conducted on a subset of participants in the trial who will be enrolled towards the end in order to assess the level of acceptability of PDMC; adaptations to health workers working practices to implement the intervention; perceptions of the feasibility of implementing PDMC through different delivery mechanisms and generate recommendations for effective implementation and job aides to support scale-up.

Effectiveness evaluation endpoints:

The primary endpoint is the proportion of children with incomplete adherence to the 9 doses of PDMC (three courses of 3-day treatments 3x3=9). Secondary endpoints include: i) incidence of all-cause and malaria-specific readmissions by the end of week 14 after discharge; ii) incidence of all-cause and malaria-specific sick-child clinic visits by 14 weeks after discharge; iii) incidence of all-cause mortality by 14 weeks after discharge.

Economic evaluation endpoints:

The primary endpoint is the incremental cost per DALY averted of alternative PDMC adherence support strategies (adherence support option A [Aa], adherence support option B [Ab]) with no adherence support (Ac), and with each other. Secondary endpoints include cost per additional child receiving a complete dose of PDMC, cost per hospital readmission averted, cost per child receiving a complete dose, cost per readmission event, cost per hospital and cost per child, and cost per child death; percentage change in budget required to deliver the intervention.

Acceptability and feasibility evaluation endpoints: i) health provider, manager and policy stakeholder acceptability of the regimen and perceptions of caregiver acceptability and adherence; ii) health provider, manager and policy stakeholder perceptions of the feasibility of each delivery strategy when implemented at scale, and adaptations to their working practices required to ensure effective implementation, and iii) caregiver and community health worker acceptability of the regimen and the alternative delivery strategies in each trial.

Follow-up procedures: Caregivers of eligible children will be approached for potential participation during hospitalization by dedicated study staff, and a consent form will be administrated near or on the day of discharge. Two nurses will be assigned to each site to oversee recruitment. Under the supervision of the study coordinator, they will schedule follow-up visits after randomisation. After consent is obtained and before discharge, household addresses will be collected, including caregivers phone contacts. The study staff will conduct a household visit to accurately identify the homes location for future visits, including GPS coordinates to facilitate future identification of households. A household questionnaire will be administered at this time including data to assess socioeconomic status. Before and during the trial, several sensitization activities will be conducted with on-site health workers, community health workers, and local community leaders (heads of villages and sub-districts) to explain the purpose of the study. Meetings with on-site health workers will also be held periodically to maintain their commitment to the trial and identify eligible children. An annual stakeholder meeting will also be held to maintain national engagement and support.

Children will be followed for 14 weeks (i.e., four weeks after the last PDMC course) through passive surveillance of clinic visits and hospitalisations. Each child will then be seen for an end-of-study visit towards the end of week 14. Children will also be visited at home for unannounced home visits one to three days from the last day of the last dose of each 3-day course of PDMC medication to assess adherence.

Sample size: A sample size of 180 participants in the control arm (c) and 180 in each of the two intervention arms (a and b), totaling 540 participants, would provide 90% power to detect a 50% reduction in the primary endpoint (proportion of children with incomplete adherence to the 9 doses of PDMC) from 36.8% in the control arm to 18.4% (RR=0.50) in any of the two intervention arms using a 1:1:1 allocation after accounting for the multiple comparisons (α = 0.025) and the correlation between participants from the same village followed by the same CHW using the very small intra-cluster correlation coefficient (ICC) value of 7.56e-0614. A total of 648 participants (216 per arm) will be recruited from the two health facilities to allow for a 15% loss to follow-up with an average of 6 participants per cluster with 36 clusters per arm selected.

Trial effectiveness analysis: Risk ratios and corresponding 95% confidence intervals will be computed to compare treatment effects using generalised linear mixed model (GLMM). Covariate-adjusted analyses for the primary endpoint will also be conducted by adding pre-specified covariates into the above unadjusted GLMM analysis to derive the adjusted RR (95% CI). The random effect for cluster will be removed if the model cannot converge. Small-sample correction will be considered given the relatively low number of clusters recruited using adjusted degrees of freedom to follow the t-distribution, rather than the normal distribution, or bootstrapping method to get valid variance estimates. A detailed study statistical analytical plan for the final analysis, that will supersede the study protocol, will be drawn up during the study at database lock.

Economic, acceptability, and feasibility evaluation analysis: Framework analysis will be used to identify factors influencing the effectiveness and scalability of each intervention delivery strategy. We will draw on multiple frameworks whereby initial coding will be based on key elements using a pre-defined PDMC implementation framework [9] and the building blocks of the health system as defined by the World Health Organization [10]. Acceptability theory will draw on Sekhon's constructs of acceptability [11] - affective attitude (general feelings about the intervention), burden (perceptions of effort needed to take part), ethicality (fit with their value system), intervention coherence (understanding of the intervention and how it works), opportunity costs (what must be given up in order to participate), perceived effectiveness (perceptions of the intervention's ability to achieve its aim), and self-efficacy (feeling that they can do what they need to do to take part) and unintended consequences.

Adverse events analysis: AE data will be collected but will be presented mainly in a descriptive way. The frequency and percentages of each event will be indicated by the intervention arm. Treatment-emergent adverse events are defined as adverse events that had an onset on or after the day of the first dose of study medication. Adverse events that have missing onset dates will be considered to be treatment-emergent. No formal statistical testing will be undertaken.

Timeframe and duration of the study: The total duration of the study is 36 months (January 2024-December 2026), including 9-12 months of study preparation (January -September 2024: protocol preparation and approvals; October -December 2024: study preparation and set-up), approximately 16-18 months of recruitment and follow-up (January 2025-June 2026) and 6-8 months of data analysis and report writing (July 2026 - December 2026).

Ethical committee and national regulatory authorities approvals will be obtained before the trial starts.

References:

1. Kwambai TK, Mori AT, Nevitt S, et al. Post-discharge morbidity and mortality in children admitted with severe anaemia and other health conditions in malaria-endemic settings in Africa: a systematic review and meta-analysis. Lancet Child Adolesc Health 2022.
2. Opoka RO, Hamre KES, Brand N, Bangirana P, Idro R, John CC. High Postdischarge Morbidity in Ugandan Children With Severe Malarial Anemia or Cerebral Malaria. J Pediatric Infect Dis Soc 2017; 6(3): e41-e8.
3. van Hensbroek MB, Jonker F, Bates I. Severe acquired anaemia in Africa: new concepts. Br J Haematol 2011; 154(6): 690-5.
4. Kwambai TK, Dhabangi A, Idro R, et al. Malaria Chemoprevention in the Postdischarge Management of Severe Anemia. N Engl J Med 2020; 383(23): 2242-54.
5. Bojang KA, Milligan PJ, Conway DJ, et al. Prevention of the recurrence of anaemia in Gambian children following discharge from hospital. PloS one 2010; 5(6): e11227.
6. Phiri K, Esan M, van Hensbroek MB, Khairallah C, Faragher B, ter Kuile FO. Intermittent preventive therapy for malaria with monthly artemether-lumefantrine for the post-discharge management of severe anaemia in children aged 4-59 months in southern Malawi: a multicentre, randomised, placebo-controlled trial. The Lancet Infectious diseases 2012; 12(3): 191-200.
7. World Health Organisation Global Malaria Programme. WHO Guidelines for malaria - 3 June 2022 (https://apps.who.int/iris/rest/bitstreams/1427681/retrieve). Geneva, 2022.
8. Nkosi-Gondwe T, Robberstad B, Mukaka M, et al. Adherence to community versus facility-based delivery of monthly malaria chemoprevention with dihydroartemisinin-piperaquine for the post-discharge management of severe anemia in Malawian children: A cluster randomized trial. PloS one 2021; 16(9): e0255769.
9. Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci 2009; 4: 50.
10. World Health Organisation. Everybodys Business: Strengthening Health Systems to Improve Health Outcomes: Framework for Action. Geneva, WHO, ISBN 978 92 4 159607 7, http://wwwwhoint/healthsystems/strategy/everybodys_businesspdf accessed 7 June 2014 2007.
11. Sekhon M, Cartwright M, Francis JJ. Acceptability of healthcare interventions: an overview of reviews and development of a theoretical framework. BMC Health Serv Res 2017; 17(1): 88

ELIGIBILITY:
Inclusion Criteria:

* Aged below 10 years of both sexes
* Hospitalised with severe anaemia or severe malaria: Initially hospitalised with haemoglobin below 5.0 g/dl or PCV below 15%, or requirement for blood transfusion for other clinical reasons on or during admission to the hospital, or severe malaria, defined as a requirement for parenteral artesunate in the opinion of the treating clinician and the presence of microscopy or RDT confirmed Plasmodium infection

Exclusion Criteria:

* Recognised specific other causes of severe anaemia (i.e., trauma, haematological malignancy, known bleeding disorders, such as haemophilia)
* Sickle cell anaemia/sickle cell disease
* Body weight below 5 kg
* HIV infection and cotrimoxazole prophylaxis are not exclusion criteria

Max Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 648 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of children with incomplete adherence to 9 doses of PDMC by the end of week 14 post-discharge | Administration of PDMC courses at 2, 6 and 10 weeks post discharge
  Adherence to the PDMC strategy: Proportion of children with incomplete adherence to 9 doses of PDMC (three courses of 3-day treatments 3x3=9) i.e. the number of children who do not receive the total of 9 doses of PDMC tablets by the end of week 14 after discharge out of the total sample size.

SECONDARY OUTCOMES:
Number of children readmitted to hospital from all-cause and malaria-specific by the end of week 14 post-discharge | 14 weeks post discharge
  Incidence of all-cause and malaria-specific readmissions by the end of week 14 after discharge, i.e. the number of children readmitted for malaria by the end of week 14 after discharge out of the total sample size.
Number of sick-child clinic visits from all-cause and malaria-specific by the end of week 14 post-discharge | 14 weeks post discharge
  Proportion of all-cause and malaria-specific sick-child clinic visits by the end of week 14 after discharge, i.e. the number of children who visit the hospital for any cause or due to malaria by the end of week 14 after discharge out of the total of sample size
Number of children who die within 14 weeks post-discharge | 14 weeks post discharge
  Incidence of all-cause mortality of children by the end of week 14 after discharge, i.e. the number of children who die within 14 weeks of discharge out of the total sample size
Number of serious adverse events following PDMC administration within 14 weeks post-discharge | 14 weeks post discharge
  Safety of PDMC strategy: Proportion of serious adverse events occurring after discharge to 14 weeks post-discharge, i.e. the number of children presenting serious adverse events by the end of week 14 after discharge out of the total sample size
Cost per Disability adjusted life years (DALY) averted for each intervention versus control arm | 14 weeks post discharge
  DALYs will be determined at the individual level and calculated based on the standard method used by the 2010 Global Burden of Disease Study (and using disability weights and life expectancies at age of death from the most recent WHO life tables). The total number of DALYs will be calculated by adding the DALYs for each individual who receives the intervention/s. The cost per DALY averted for each intervention will be compared against published country-specific willingness-to-pay thresholds to assess cost-effectiveness
Stakeholder perceptions of the feasibility on the delivery strategy with adherence supports | Within 6 month following the benning of trial
  Health providers, managers, health community workers, and policy stakeholders' perceptions regarding the feasibility of the delivery strategy and adherence support by assessing barriers and constraints through focus group discussions and key in-depth interviews.
Stakeholder acceptability of the regimen of the PDMC strategy and perception of caregiver acceptability and adherence | Within 6 month following the benning of trial
  Health providers, managers, health community workers, and policy stakeholders acceptability regarding the acceptability of the regimen and the perception of the caregivers acceptability and adherence. Acceptability theory will draw on Sekhon's constructs of acceptability - - affective attitude (general feelings about the intervention), burden (perceptions of effort needed to take part), ethicality (fit with their value system), intervention coherence (understanding of the intervention and how it works), opportunity costs (what must be given up in order to participate), perceived effectiveness (perceptions of the intervention's ability to achieve its aim), and self-efficacy (feeling that they can do what they need to do to take part) and unintended consequences.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Hill, MSc, PhD, Principal Investigator — Liverpool School of Tropical Medicine
Locations (2):
- Benin (2):
  - Goho Departmental Hospital Centre, Abomey
  - Centre Hospitalier Universitaire de la Mere et de l'Enfant Lagune (CHU-MEL), Cotonou

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be shared once the publication is accepted by a journal
Access Criteria: Applications to access data are assessed as per the choice of the data contributor, either by:
  1. An independent IDDO Data Access Committee (DAC)
  2. A contributor-controlled process - where the data contributor assesses each data access application that requests the re-use of their data
URL: https://www.iddo.org/data-sharing/contributing-data

REFERENCES:
- [Background] Hill J; PDMC Saves Lives Consortium. Implementation of post-discharge malaria chemoprevention (PDMC) in Benin, Kenya, Malawi, and Uganda: stakeholder engagement meeting report. Malar J. 2024 Mar 27;23(1):89. doi: 10.1186/s12936-023-04810-0. PMID 38539181